CLINICAL TRIAL: NCT00477295
Title: A Randomized, Multi-centre, Double-blind Study, to Compare the Efficacy and Safety of Zonisamide and Carbamazepine as Monotherapy, in Newly Diagnosed Partial Epilepsy
Brief Title: A Double-blind Study to Compare the Efficacy and Safety of Zonisamide and Carbamazepine as Monotherapy, in Newly Diagnosed Partial Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2090-E044-310; 2006-000156-40 (EudraCT Number)
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide; Carbamazepine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Zonisamide (Active Comparator)
  Interventions: Drug: Zonisamide
- Carbamazepine (Active Comparator)
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Zonisamide — Week 1 and 2 either 100mg zonisamide or 200 mg carbamazepine Week 3 and 4 either 200mg zonisamide or 4800 mg carbamazepine Week 5 and 6 either 300mg zonisamide or 600 mg carbamazepine; this dose then to be maintained unless a subject has a seizure more than two weeks post a dose increase.
  Other Names: Zonegran
  Arms: Zonisamide
Drug: Carbamazepine — Week 1 and 2 either 100mg zonisamide or 200 mg carbamazepine Week 3 and 4 either 200mg zonisamide or 4800 mg carbamazepine Week 5 and 6 either 300mg zonisamide or 600 mg carbamazepine; this dose then to be maintained unless a subject has a seizure more than two weeks post a dose increase.
  Arms: Carbamazepine

SUMMARY:
This is a two-arm, randomized, double-blind, non-inferiority study using a flexible dosing regime to allow optimal zonisamide or carbamazepine therapy for individual subjects. Assessment of eligibility will take place at the Screening Visit. The subjects will be randomized to either the carbamazepine or zonisamide arm at the Randomization Visit (T1). T1 must occur as soon as possible (and at least within 14 days) of the Screening Visit in order to optimize subject care.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects will be eligible for the study if they meet all of the following inclusion criteria:

1. Male or female subjects, 18 to 75 years of age inclusive.
2. Subjects with untreated, newly diagnosed epilepsy having at least two well documented, unprovoked, clinically evaluated and classified partial seizures (with or without secondary generalization) or generalized tonic-clonic seizures (without clear focal origin) within 12 months of the Screening Visit, of which at least one seizure occurred within three months of the Screening Visit (> one seizure within a 24 hour period will be counted as one seizure).
3. Subjects will either have had no previous use of an AED, or treatment with one AED for a maximum duration of two weeks before the Randomization Visit (T1).
4. Subjects have a documented electroencephalogram (EEG) within 12 months of the Screening Visit, compatible with localization-related epilepsy (to exclude primary generalized epilepsy).
5. Subjects have a documented computed axial tomography (CAT) scan or magnetic resonance imaging (MRI) scan confirming the absence of a progressive neurological lesion within 12 months of the Screening Visit.
6. Female subjects without childbearing potential (two years post-menopausal, bilateral oophorectomy or tubal ligation, complete hysterectomy) are eligible. Female subjects with childbearing potential must not be pregnant as confirmed by a negative pregnancy test at screening and randomization, must not be lactating and must be using a medically acceptable form of contraception, for the duration of the study and for one month following discontinuation of the study drug. Medically acceptable contraception is defined here as oral contraception pill with at least 50 micrograms ethinylestradiol per intake, contraceptive injections and implants, or intrauterine device in place for at least three months.
7. Subjects who are able and willing to follow investigational study procedures, maintain a seizure diary, and report AEs.
8. Subjects who are able and willing to give written informed consent.

EXCLUSION CRITERIA:

Subjects who meet any of the following exclusion criteria will not be eligible for the study:

1. Subjects have a history of clinical investigations, including EEG data, that are suggestive of idiopathic generalised epilepsy as defined by the International League Against Epilepsy (ILAE).
2. Subjects with a history of absence, myoclonic, clonic, tonic, or atonic seizures.
3. Subjects have a history of status epilepticus, and/or non-epileptic seizures (e.g., metabolic, pseudo-seizures).
4. Subjects have experienced seizures relating to drugs, alcohol, acute medical illness, mental retardation, or subjects with situation-related seizures.
5. Subjects have progressive encephalopathy or findings consistent with progressive CNS disease or lesion (e.g. infection, demyelination, or tumour).
6. Subjects have a history of a significant or currently uncontrolled disease that will interfere with the conduct of this study or the assessment of safety and efficacy of the study drug.
7. Subjects have been previously treated with carbamazepine or zonisamide.
8. Subjects have received an investigational drug or device in the three months prior to the Screening Visit.
9. Subjects have a known hypersensitivity to sulfonamides, dibenzazepine derivatives, or tricyclic antidepressants.
10. Subjects have a history of bone marrow depression, low platelet count or other blood dyscrasia.
11. Subjects have a history of acute intermittent porphyria.
12. Subjects have a history of renal disorder (serum creatinine level of > 135 Ã¬mol / l (1.5 mg/dL at the Screening Visit), hepatic disorder or clinically significant abnormal liver function tests; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2 times the upper normal limit.
13. Subjects have a body weight of less than 40 kg.
14. Subjects have a history of progressive malignancy within the previous 5 years (excluding a history of non-metastasized and adequately treated cutaneous squamous cell carcinoma).
15. Subjects have a history of psychiatric illness or mood disorder requiring electro-convulsive or drug therapy within the previous 6 months which is considered uncontrolled; a history of suicide attempt; alcohol or drug abuse; chronic treatment with benzodiazepines or barbiturates.
16. Subjects are currently taking carbonic anhydrase inhibitors.
17. Subjects have a history of pancreatitis, nephrolithiasis or hypercalcuria, clinically significant laboratory or electro-cardiographic abnormalities, or uncontrolled hypertension.
18. Subjects are currently taking mono-amine oxidase inhibitors (MAOIs) or any other excluded medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Segieth, Study Director — Eisai Limited
Locations (79):
- Australia (8):
  - Camperdown
  - Clayton
  - Fitzroy
  - Flinders
  - Heidelberg West
  - Parkville
  - Queensland
  - Wellington
- Aalborg, Denmark
- France (4):
  - Béthune
  - Dijon
  - Paris
  - Saint-Etienne
- Germany (6):
  - Berlin
  - Bochum
  - Düsseldorf
  - Munich
  - Schwerin
  - Westerstede
- Greece (2):
  - Athens
  - Thessaloniki
- Hungary (6):
  - Budapest
  - Debrecen
  - Gyula
  - Hódmezővásárhely
  - Nyregyhaza
  - Zalaegerszeg-Pozva
- India (6):
  - Bangalore
  - Hyderabad
  - Koturpuram
  - Madurai
  - New Delhi
  - Pune
- Italy (4):
  - Milan
  - Monza
  - Orbassano
  - Rome
- Poland (9):
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Sosnowiec
  - Szcecin
  - Warsaw
- Russia (5):
  - Kaliningrad
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Yaroslavl
- Serbia (4):
  - Belgrade
  - Niš
  - Novi Sad
  - Subotica
- Slovakia (6):
  - Bratislava
  - Bratslava
  - Brezno
  - Nové Zámky
  - Vranov nad Topľou
  - Žilina
- Sandton, South Africa
- South Korea (3):
  - Anyang
  - Seoul
  - Wŏnju
- Spain (7):
  - Alicante
  - Bacelona
  - Barcelona
  - Madrid
  - Málaga
  - Oviedo
  - Seville
- Sweden (2):
  - Gothenburg
  - Lund
- Taiwan (2):
  - Changhua
  - Yongkang District
- United Kingdom (3):
  - Bristol
  - Liverpool
  - Treliske

REFERENCES:
- [Derived] Baulac M, Brodie MJ, Patten A, Segieth J, Giorgi L. Efficacy and tolerability of zonisamide versus controlled-release carbamazepine for newly diagnosed partial epilepsy: a phase 3, randomised, double-blind, non-inferiority trial. Lancet Neurol. 2012 Jul;11(7):579-88. doi: 10.1016/S1474-4422(12)70105-9. Epub 2012 Jun 8. PMID 22683226

RESULTS

PARTICIPANT FLOW:
Groups:
- Zonisamide: The starting dose in this arm was zonisamide 100mg daily. The dose during the Titration Period (4 weeks) ranged from 100 to 200mg daily. During the Flexible Dosing Period (FDP), the subjects were given doses ranging from 300 to 500mg daily or if they could not tolerate that dose, were allowed one down-titration or were withdrawn. If the subjects remained seizure-free for 26 weeks by the end of FDP (the subject was allowed 3 chances to achieve this), they entered the Maintenance Period (26 weeks), where they remained on the same dose they were taking at the end of the FDP.
- Carbamazepine: The starting dose in this arm was carbamazepine 200mg daily. The dose during the Titration Period (4 weeks) ranged from 200 to 400mg daily. During the Flexible Dosing Period (FDP), the subjects were given doses ranging from 600 to 1200mg daily or if they could not tolerate that dose, were allowed one down-titration or were withdrawn. If the subjects remained seizure-free for 26 weeks by the end of FDP (the subject was allowed 3 chances to achieve this), they entered the Maintenance Period (26 weeks), where they remained on the same dose they were taking at the end of the FDP.
Period: Overall Study
Arm/Group | Zonisamide | Carbamazepine
Started | 282 | 301
Completed | 161 | 192
Not Completed | 121 | 109
Not completed — Adverse Event | 31 | 35
Not completed — Withdrawal by Subject | 35 | 24
Not completed — Lack of Efficacy | 23 | 23
Not completed — Protocol Violation | 3 | 8
Not completed — Physician Decision | 4 | 5
Not completed — Lost to Follow-up | 21 | 11
Not completed — Other | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Zonisamide: The starting dose in this arm was zonisamide 100mg daily. The dose during the Titration Period (4 weeks) ranged from 100 to 200mg daily. During the Flexible Dosing Period (FDP), the subjects were given doses ranging from 300 to 500mg daily or if they could not tolerate that dose, were allowed one down-titration or were withdrawn. If the subjects remained seizure-free for 26 weeks by the end of FDP(the subject was allowed 3 chances to achieve this), they entered the Maintenance Period (26 weeks), where they remained on the same dose they were taking at the end of the FDP.
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Carbamazepine | Total
Number analyzed (Participants) | 281 | 300 | 581
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety Population.
  years | 37.1 (16.33) | 35.6 (15.50) | 36.4 (15.91)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population: All randomized subjects who received at least one dose of study medication.
  Participants
    Female | 107 | 128 | 235
    Male | 174 | 172 | 346

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Seizure Freedom for 26-weeks During the Maintenance Phase
Description: A subject achieved a 26-week seizure-free period if they were free of all seizures, regardless of seizure type, for 26 weeks while receiving the same dose. The occurrence of seizures was documented in the seizure diary, which was maintained by the subject and reviewed at each following visit.
Time Frame: Week 31 through Week 109
Population: Per Protocol Population: All randomized subjects who received at least one dose of study medication and who had no major protocol violations.
Measure: Number; unit: Percentage of Participants
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 223 | 233
Percentage of Participants | 79.4 | 83.7

2. Secondary Outcome: Percentage of Participants Who Experienced Seizure Freedom for 12-months During the FDP and Maintenance Period
Description: A subject achieved a 12-month seizure-free period if they were free of all seizures, regardless of seizure type, for 12 months while receiving the same dose. The occurrence of seizures was documented in the seizure diary, which was maintained by the subject and reviewed at each following visit.
Time Frame: Week 5 through Week 109
Population: Per Protocol Population. N=number of subjects with evaluable data.
Measure: Number; unit: Percentage of participants
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 216 | 229
Percentage of participants | 67.6 | 74.7

3. Secondary Outcome: Analysis of Time to Drop Out Due to an Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a subject and does not necessarily have a causal relationship with the medicinal product. Adverse events were identified by: any unfavorable or unintended sign, symptom or disease temporarily associated with the use of a medicinal product; any new disease or exacerbation of an existing disease; any deterioration in nonprotocol-required measurements of laboratory values or other clinical test; and recurrence of an intermittent medical condition not present at Baseline.
Time Frame: Week 1 through Week 109
Population: Per Protocol Population
Measure: Median (Standard Error); unit: Median Days
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 223 | 233
Median Days | NA (NA) — Please note that this is reported as 'Not Calculable' due to insufficient events. | NA (NA) — Please note that this is reported as 'Not Calculable' due to insufficient events.

4. Secondary Outcome: Analysis of Time to Drop Out Due to Lack of Efficacy
Description: Lack of efficacy was evaluated by the subject and on the basis of whether zonisamide and carbamazepine gave the subject at least a 26-week seizure free rate. The subject could withdraw at any time due to lack of efficacy.
Time Frame: Week 1 through Week 109
Population: Per Protocol Population
Measure: Median (Standard Error); unit: Median Days
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 223 | 233
Median Days | 722 (NA) — Please note that this is reported as 'Not Calculable' due to insufficient events. | NA (NA) — Please note that this is reported as 'Not Calculable' due to insufficient events.

5. Secondary Outcome: Time to 6-months Seizure Freedom
Description: A subject achieved a 6-months seizure-free period if they were free of all seizures, regardless of seizure type, for 6-months while receiving the same dose. The occurrence of seizures was documented in the seizure diary, which was maintained by the subject and reviewed at each following visit.
Time Frame: Week 5 through Week 83
Population: Intent-to-Treat (ITT) Population - randomized subjects who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 281 | 300
Days | 222.7 (49.78) | 220.4 (46.31)

6. Secondary Outcome: Time to 12-months Seizure Freedom
Description: A subject achieved a 12-month seizure-free period if they were free of all seizures, regardless of seizure type, for 12-months while receiving the same dose. The occurrence of seizures was documented in the seizure diary, which was maintained by the subject and reviewed at each following visit.
Time Frame: Week 5 through Week 83
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 281 | 300
Days | 399.3 (55.03) | 395.6 (42.19)

7. Secondary Outcome: Change From Baseline in Total ABNAS Score at Maintenance Period Visit 1
Description: The Aldenkamp-Baker Neuropsychological Assessment Scale(ABNAS) is a subject based questionnaire to measure subjective perceived drug-related cognitive impairments. The ABNAS measured seven critical domains of cognition(tiredness/fatigue,hyperexcitability, slowing(mental and motor),memory impairment,attention disorders,impairment of motor coordination, and language disorders). The total score ranged from 0 to 72, with a higher score reflecting a high level of problems.
Time Frame: Baseline and Maintenance Period Visit 1 (Week 31 to Week 83)
Population: Intent-to-Treat Population: All randomized subjects who received at least one dose of study medication. This was measured using Observed Case (OC).
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 281 | 300
Scores on a Scale | 1.6 (15.43) | -0.1 (12.71)

8. Secondary Outcome: Change From Baseline in Bond and Lader VAS Mood Sub-Scores at Maintenance Period Visit 1
Description: The Bond-Lader Visual Analogue Scale (VAS) is made up of 16 pairs of alternative descriptors of mood and attention at either end of a 10 cm line.
  Subjects were asked to rate their feelings at the time of assessment by indicating the point on the line which best represent their mood. Each item was scored by measuring the position relative to the left hand end of the line and levels of anxiety, sedation, and dysphoria were then calculated from the combined scores of selected items. The scores ranged from 0 to 100, with a high score reflecting a high level of anxiety, sedation or dysphoria.
Time Frame: Baseline and Maintenance Period Visit 1 (Week 31 to Week 83)
Population: Intent-to-Treat Population. This was measured using Observed Case (OC).
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 281 | 300
Scores on a Scale
  Anxiety | -2.036 (23.6120) | -1.993 (26.1087)
  Sedation | -0.475 (21.7476) | -1.362 (18.0103)
  Dysphoria | -1.930 (21.7585) | -3.833 (19.7824)

9. Secondary Outcome: Change From Baseline in QOLIE-31-P Overall Score at Maintenance Period Visit 1
Description: The Quality of Life in Epilepsy - Problems(QOLIE-31-P) was completed by the patient and contained 30 items covering seven subscales(seizure worry, overall
  Quality of Life (QOL),emotional well-being,energy-fatigue, cognition,medication effects and social function) and one item covering health status. It also included seven items addressing overall distress related to each subscale, an item addressing the relative importance of each subscale topic, and an item addressing perception of overall change in QOL at the end of the study. A high score reflects a good QOL. The following scale range is a sample of 1 of the 7 of the subscales:
  10 (Best possible quality of life) - 0 (Worst possible quality of life);
  Rand Corporation QOLIE-31 Scoring Manual was used. The QOLIE-31 overall score is calculated by summing the product of each scale score times its weight and summing overall all scales.
Time Frame: Baseline and Maintenance Period Visit 1 (Week 31 to Week 83)
Population: Intent-to-Treat Population. This was measured using Observed Case (OC).
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 281 | 300
Scores on a Scale | 4.474 (15.2838) | 6.090 (13.2861)

10. Secondary Outcome: Change From Baseline in SF-36 Aggregate Mental and Physical Component Score at Maintenance Period Visit 1
Description: The Short Form 36 Health and Well-Being Questionnaire (SF-36) is a 36-item generic health related QOL instrument covering the following domains: physical functioning, role-physical,bodily pain, general health, social functioning,role-emotional, mental health, and vitality. It yields a profile of eight scores, one for each domain, and physical and mental health summary measures. Each domain is described by a score ranging from 0 to 100, for a range of total possible scoes of 0-400 for physical and 0-400 for mental. An increase represents an improvement, whereas a decrease reflects a worsening.
Time Frame: Baseline and Maintenance Period Visit 1 (Week 31 to Week 83)
Population: Intent-to-Treat Population. This was measured using Observed Case (OC).
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 281 | 300
Scores on a Scale
  Aggregate Mental Component Score | 1.027 (10.9124) | 2.495 (10.5310)
  Aggregate Physical Component Score | 1.895 (7.6287) | 2.041 (6.2613)

11. Secondary Outcome: Percentage of Participants With EQ-5D Scores at Maintenance Period Visit 1
Description: The European Quality of Life Group 5-Dimension Self-Report Questionnaire (EQ-5D) is a preference based generic health related quality of life (HRQoL) instrument which classifies health states across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain has three levels, they are (1) no problems, (2) some problems, (3) extreme problems. The percentages shown are calculated from the number of subjects at that visit with non-missing data for that score.
Time Frame: Week 31 through Week 83
Population: Intent-to-Treat Population. This was measured using Observed Case (OC). The percentages shown are calculated from the number of subjects at that visit with non-missing data for that score (n=174,196).
Measure: Number; unit: Percentage of Participants
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 174 | 196
Percentage of Participants
  Mobility: No problems | 90.8 | 86.7
  Mobility: Some problems | 8.7 | 12.9
  Mobility: Confined to Bed | 0.5 | 0.5
  Self-Care:No problems | 96.7 | 97.6
  Self-Care: Some problems | 2.7 | 2.4
  Self-Care: Unable to wash or dress | 0.5 | 0.0
  Usual Activities: No problems | 89.1 | 84.8
  Usual Activities: Some problems | 9.8 | 15.2
  Usual Activities: Unable to perform | 1.1 | 0.0
  Pain/Discomfort: None | 75.5 | 73.2
  Pain/Discomfort: Moderate | 22.3 | 25.4
  Pain/Discomfort: Extreme | 2.2 | 1.4
  Anxiety/Depression: None | 64.3 | 62.9
  Anxiety/Depression: Moderate | 31.3 | 34.8
  Anxiety/Depression: Extreme | 4.4 | 2.4

ADVERSE EVENTS:
Time Frame: A Treatment-Emergent Adverse Event (TEAE) is an Adverse Event (AE) with a start date on or after Day 1 and within 15 days of last dose, including AEs with missing start dates, for up to 116 weeks.
Description: For each AE category, a subject with two or more adverse events in that category is only counted once.
Arm/Group | Zonisamide | Carbamazepine
Serious Adverse Events (participants affected / at risk) | 15/281 | 17/300
Other Adverse Events (participants affected / at risk) | 72/281 | 69/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide (N=281) | Carbamazepine (N=300)
Partial seizures with secondary generalization (Nervous system disorders) | 0 | 4
Complex partial seizures (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Ischemic stroke (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Subarachnoid hemorrahage (Nervous system disorders) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Sinusitis bacterial (Infections and infestations) | 0 | 1
Typhoid fever (Infections and infestations) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Death (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide (N=281) | Carbamazepine (N=300)
headache (Nervous system disorders) | 29 | 37
somnolence (Nervous system disorders) | 17 | 23
dizziness (Nervous system disorders) | 11 | 23
weight decreased (Investigations) | 19 | 0
decreased appetite (Metabolism and nutrition disorders) | 22 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No